CLINICAL TRIAL: NCT00475202
Title: Hyperbaric Oxygen Therapy and Angiogenesis in Diabetic Patients With Foot Ulcers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 6106
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Last update posted 2007-05-21 (Estimated); Status verified 2007-05

CONDITIONS: Diabetic Foot Ulcers; Hyperbaric Therapy; Angiogenesis
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Diabetic foot ulcers are a major cause of morbidity and mortality, accounting for approximately two-thirds of all non-traumatic amputations performed in the United States. The cost of foot ulcers in diabetic patients averages almost $28,000 for the two years after diagnosis of the ulcer. Hyperbaric oxygen (HBO) serves as primary or adjunctive therapy for a diverse range of medical conditions. HBO also has been used as an adjunct to antibiotics, debridement, and revascularization in the therapy of chronic, nonhealing wounds associated with diabetes or non-diabetic vascular insufficiency.

The aim of the study is to assess whether hyperoxia induced angiogenesis in diabetic patients with foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older, with type II diabetes suffering from foot ulcers admitted to the Institute of Hyperbaric Medicine and Wound Care Clinic at Assaf Harofeh Medical Center (Israel)

Exclusion Criteria:

* Patients having chest pathology incompatible with pressure changes, inner ear disease, or suffering from claustrophobia, will be excluded from the study. Patients with significant macrovascular disease, defined as obstruction of more than 50% in the femoral or the popliteal arteries, will also be excluded from the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Albert Rabinovitz, MD, Principal Investigator — Assaf-Harofeh Medical Center; Efrati Shai, MD, Study Chair — Assaf-Harofeh Medical Center
Locations (1):
- Institute of Hyperbaric Medicine and Wound Care Clinic at Assaf Harofeh Medical Center, Ẕerifin, Israel